CLINICAL TRIAL: NCT04668183
Title: Ultrasound-guided Pudendal Nerve Block Versus Ultrasound-guided Dorsal Penile Nerve Block for Pediatric Distal Hypospadias Surgery
Brief Title: Ultrasound-guided PNB and DPNB for Pediatric Distal Hypospadias Surgery
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Volkan Ozen, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: 1457
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Regional Anesthesia; Hypospadias
Keywords: Postoperative pain; Ultrasound; Dorsal penile nerve block; Pudendal nerve block; Hypospadias
MeSH Terms: conditions — Hypospadias; Pain, Postoperative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pudendal Nerve Block: Linear ultrasound probe and the sacral hiatus at the sacral cornu level was visualized using an out-of-plane transverse view at 5-10 megahertz . The linear probe was then rotated 90 degrees and placed longitudinally in the midline to evaluate the sacral cornus, sacrococcygeal ligament and sacral bone.
  Interventions: Procedure: Pudendal nerve block group
- Dorsal Penile Nerve Block: Ultrasound (US) guided dorsal penile nerve block with in plane technique was done. Half of the total 0.2 ml/kg dose of 0.25% bupivacaine was administered while observing its distribution with US. The same procedure was then repeated on the other side of the penis.
  Interventions: Procedure: Dorsal penile nerve block group

INTERVENTIONS:
Procedure: Pudendal nerve block group — A 22 Gauge 50 mm insulated needle was then introduced in the anterior-posterior direction at the middle of the ultrasound probe's superior edge with an out-of-plane approach and using an inclination of 15° in the sagittal plane. The needle tip's position was identified by direct visualization using the movement of adjacent anatomical structures.
  Groups: Pudendal Nerve Block
Procedure: Dorsal penile nerve block group — Half of the total 0.2 ml/kg dose of 0.25% bupivacaine was administered while observing its distribution with US. The same procedure was then repeated on the other side of the penis.
  Groups: Dorsal Penile Nerve Block

SUMMARY:
Hypospadias repair is a urological surgical operation that is very painful in the postoperative period and requires long-term analgesia. A dorsal penial nerve block (DPNB) and pudendal nerve block (PNB), which are regional anesthesia techniques for this operation, are used to provide postoperative analgesia.

DETAILED DESCRIPTION:
The regional anesthesia techniques used for postoperative analgesia in hypospadias repair include the peripheral nerve blocks of pudendal nerve block (PNB) and dorsal penile nerve block (DPNB). Ultrasound (US) has recently become increasingly popular in regional anesthesia practice and is used to aid these two peripheral nerve block applications in various pediatric urological procedures. US-guided DPNB has been shown to provide effective and long-term analgesia when compared to caudal epidural block in a recent study on hypospadias surgery in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged between 1-7 years
* American Society of Anesthesiologists (ASA) I-II group
* Distal hypospadias surgery
* Able to communicate in Turkish
* Willing to participate to the study (parents and children)

Exclusion Criteria:

* Less than 1 or more than 7 years of age
* A neurological deficit, bleeding diathesis, or a history of local anesthetic allergy; an infection or redness in the injection area, congenital low back anomaly, liver disorder, a psychiatric disorder, mental retardation, or communication problems detected during examination
* Unwilling to to participate to the study ((parents or children)

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study was conducted with children who underwent hypospadias surgery at a training and research hospital in Istanbul, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Time of Postoperative analgesic requirement | Up to 24 hours
  It was assessed six times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 1st, 2nd, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse. Paracetamol was administered IV at a dose of 10 mg/kg if the scale score was 7 or higher.

SECONDARY OUTCOMES:
Level of Postoperative pain | Up to 24 hours]
  It was assessed six times after the operation with Children's Hospital Eastern Ontario Pain Scale. The lowest scale score is 4 points and the highest 13 points. Significant pain behavior for Children's Hospital Eastern Ontario Pain Scale has been identified as 7 points or more. Following transfer from the recovery unit to the ward, the 1st, 2nd, 6th, 12th and 24th hour pain levels were evaluated by the ward nurse
Rate of Postoperative complications | Up to 24 hours
  The presence of penile edema or an injection site ecchymosis or hematoma was evaluated by an anesthesiologist blinded to the study groups postoperatively (at 30 minutes and 1, 2, 6, 12, 18 and 24 hours).
Level of Parent satisfaction | Up to 24 hours
  The parents were asked about their satisfaction with the child's comfort and activity level [1, unsatisfied; 2, satisfied (good); 3, absolutely satisfied (excellent)] at the 24-hour follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Ozen, MD, Study Director — Prof. Dr. Cemil Tascıoglu City Hospital, Istanbul, Şişli, Turkey, 34384
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozen V, Yigit D. Caudal epidural block versus ultrasound-guided dorsal penile nerve block for pediatric distal hypospadias surgery: A prospective, observational study. J Pediatr Urol. 2020 Aug;16(4):438.e1-438.e8. doi: 10.1016/j.jpurol.2020.05.009. Epub 2020 May 20. PMID 32507565
- [Background] Alizadeh F, Heydari SM, Nejadgashti R. Effectiveness of caudal epidural block on interaoperative blood loss during hypospadias repair: A randomized clinical trial. J Pediatr Urol. 2018 Oct;14(5):420.e1-420.e5. doi: 10.1016/j.jpurol.2018.03.025. Epub 2018 May 21. PMID 29858133
- [Background] Saavedra-Belaunde JA, Soto-Aviles O, Jorge J, Escudero K, Vazquez-Cruz M, Perez-Brayfield M. Can regional anesthesia have an effect on surgical outcomes in patients undergoing distal hypospadia surgery? J Pediatr Urol. 2017 Feb;13(1):45.e1-45.e4. doi: 10.1016/j.jpurol.2016.09.011. Epub 2016 Oct 26. PMID 27956108